CLINICAL TRIAL: NCT04290832
Title: Developing and Testing Interventions to Address Use of Conscientious Objection to Deny Women's Access to Abortion Care in Mexico and South Africa
Brief Title: Developing and Testing Interventions to Address Conscientious Objection to Abortion Care in Mexico and South Africa
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped prematurely due to the COVID-19 pandemic
Sponsor: Ipas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TIE_2020_01
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Abortion, Induced; Abortion, Incomplete
MeSH Terms: conditions — Abortion, Incomplete

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CO intervention (Experimental): South Africa: All health facility staff working in facilities assigned to the intervention arm receive standard Ipas support (including monitoring of abortion service provision and support to Ipas-trained abortion providers) plus the CO intervention.
  Mexico: Doctors/anyone eligible to be an abortion provider working in facilities assigned to the intervention arm receive the CO intervention.
  Interventions: Behavioral: CO Intervention
- Control (No Intervention): South Africa: All health facility staff working in facilities assigned to the control arm receive standard Ipas support (including monitoring of abortion service provision and support to Ipas-trained abortion providers).
  Mexico: No intervention

INTERVENTIONS:
Behavioral: CO Intervention — South Africa: Values clarification and attitude transformation (VCAT) workshop with conscientious objection content, debrief session(s) with termination of pregnancy (TOP) providers to give them an opportunity to share concerns/challenges, meeting(s) with facility mangers to facilitate continued support and provision of TOP care
  Mexico: Training on abortion and conscientious objection law, posters on law, offer of legal assistance for abortion providers, scholarship to attend conference awarded on basis of quality of abortion care
  Arms: CO intervention

SUMMARY:
The primary purpose of this research is to develop strategies and interventions to mitigate the impact of conscientious objection on women's access to safe abortion care in Mexico and South Africa using a user-centered design approach and test the feasibility and effectiveness of these interventions.

DETAILED DESCRIPTION:
Conscientious objection (CO) is emerging as a growing barrier to abortion care, and evidence suggests that it is being incorrectly used as a justification for public sector medical providers and institutions to exempt themselves from their duties to provide essential reproductive health services for women. Given this, it is essential to better understand and address this misuse of CO and find ways to improve women's access to safe abortion services to prevent them from using unsafe methods which risk their health and lives.

This study will conduct formative research to more fully understand the problem of CO in Mexico and South Africa and use these findings to develop interventions and strategies to mitigate the impact of CO on women's access to safe abortion care using a user-centered design approach. Rapid randomized controlled trials will then be used to assess effectiveness of the interventions. The specific aims of this study are:

1. Improve our understanding of CO and its impact on access and quality of abortion care from providers' and facility mangers' perspectives in Mexico, and South Africa.
2. Develop strategies and interventions to mitigate the impact of CO on women's access to safe abortion care. Using the data collected, a multi-disciplinary Innovation Team will develop strategies and interventions to respond to the challenges posed by CO using a user-centered design approach.
3. Rapid-test intervention prototypes. We will test selected strategies (prototypes) in Mexico, and South Africa with assessments to determine successes, and the feasibility of scaling up these approaches.

ELIGIBILITY:
South Africa

Inclusion Criteria:

* All staff currently working in selected health facilities
* Able to provide informed consent

Exclusion Criteria:

* Unable to provide informed consent

Mexico

Inclusion Criteria:

* Doctors/anyone eligible to be an abortion provider working in selected health facilities
* Able to provide informed consent

Exclusion Criteria:

* Unable to provide informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Behavior making it easier for women to access abortion care | Past 30 days
  Proportion of health facility staff exhibiting at least one behavior to make it easier for women to access abortion care (e.g. helped a woman find the abortion care unit, provided positive support to a woman seeking abortion care, gave accurate information to a woman seeking abortion care, etc.).
Behavior making it more difficult for women to access abortion care | Past 30 days
  Proportion of health facility staff exhibiting at least one behavior to make it more difficult for women to access abortion care (e.g. gave incorrect directions to a woman seeking abortion care, told a woman abortion services were not available at the facility, tried to convince a woman that she should not have an abortion, etc.).
Intention to provide abortion service, referral, or information | Next few days
  Proportion of health facility staff reporting they would provide abortion service, referral or information to women seeking abortion care in their health unit in the next few days if needed.

SECONDARY OUTCOMES:
Interest in attending an abortion care training | Assessed at baseline and at 30-day follow-up
  Proportion of providers (doctors, nurses, or midwives) reporting being interested in attending an abortion care training.
Stigmatizing Attitudes Beliefs and Actions Scale (SABAS) score | Assessed at baseline and at 30-day follow-up
  Average Stigmatizing Attitudes Beliefs and Actions Scale (SABAS) score. The SABAS is a tool designed to measure abortion stigma at the individual and community level, ranging from a minimum of 18 to a maximum of 90. A higher score represents more stigmatizing attitudes and beliefs about women who have an abortion (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Erin Pearson, PhD, MPH, Principal Investigator — Ipas
Locations (2):
- Ipas Central America and Mexico, Mexico City, Mexico
- Ipas South Africa, Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jim A, Magwentshu M, Menzel J, Kung SA, August SA, van Rooyen J, Chingwende R, Pearson E. Stigma towards women requesting abortion and association with health facility staff facilitation and obstruction of abortion care in South Africa. Front Glob Womens Health. 2023 Jun 15;4:1142638. doi: 10.3389/fgwh.2023.1142638. eCollection 2023. PMID 37396569